CLINICAL TRIAL: NCT02550951
Title: Utility of Magnetic Resonance Lymphangiography in Postoperative Follow-up of Lymphedema: Comparison With Lymphoscintigraphy
Brief Title: Utility of MR Lymphangiography in Postoperative Follow-up of Lymphedema: Comparison With Lymphoscintigraphy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung Hong Choi, SeoulNUH, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D-1408-124-607
Record Dates: First submitted 2015-09-03; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pre-operation Lymphedema (Experimental): before magnetic resonance imaging(MRI), GADOVIST PFS [Bayer Korea] 7.5mL and local anesthetics 0.5m L mixed. and then 24 gauge needle using about 1 mL by the first , and second , the third the space between the toes intradermal injection , and then about 1-2 minutes , and massage the injection site, and Acquiring an image(coronal T1-weighted three-dimensional gradient-echo sequence) of the foot from a range including up to the pelvis from the comparison with lymphoscintigraphy
  Interventions: Procedure: lymphangiography
- post-operation Lymphedema (Experimental): before magnetic resonance imaging(MRI), GADOVIST PFS [Bayer Korea] 7.5mL and local anesthetics 0.5m L mixed. and then 24 gauge needle using about 1 mL by the first , and second , the third the space between the toes intradermal injection , and then about 1-2 minutes , and massage the injection site, and Acquiring an image(coronal T1-weighted three-dimensional gradient-echo sequence) of the foot from a range including up to the pelvis from the comparison with lymphoscintigraphy
  Interventions: Procedure: lymphangiography

INTERVENTIONS:
Procedure: lymphangiography

SUMMARY:
Its usefulness in implementing magnetic resonance angiography for postoperative follow-up of lymph lymphedema should try to evaluate and compare lymphoscintigraphy.

DETAILED DESCRIPTION:
Surgical methods include " surgical procedure to make a good lymphatic drain 'and' surgical resection with lymph tissue swelling , significant that two of lymphedema .In recent years, began receiving the spotlight this former method using micro-surgery , inde essential that in order to increase the success rate of these micro-surgery accurately assess the structural abnormalities of preoperative lymphatic and establishing the surgical plan , the primary diagnostic imaging examination of existing lymphedema Since the nuclear medicine examination as to obtain an accurate anatomical information it is also ideal for imaging in the preoperative assessment of lymphedema is precisely that you can not .

In contrast magnetic resonance lymphangiography recently developed a new magnetic resonance imaging techniques that many advantages in precision assessment of lymphedema patients.

First, there are high spatial resolution magnetic resonance lymphangiography through the lymphatic vessels to obtain the correct anatomical information .

Second, magnetic resonance lymphangiography is provide not only information about the functional status of the lymphatic anatomical information .

Third, the magnetic resonance lymphangiography minimally invasive techniques , without exposure to radiation , is relatively easy and safe , that there is a great advantage of being able to diagnose the structural and functional at the same time or later in lymphatic vessels.

The magnetic resonance lymphangiography via the lymphatic advantage given also helps to establish a specific treatment plan , as well as accurate preoperative diagnosis of lymphedema that may contribute to enhance the success of micro-surgery.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years of age
* Patients underwent preoperative and receive magnetic resonance lymphangiography and Lymphoscintigraphy At the postoperative 3 months

Exclusion Criteria:

* Patients with a history of adverse effects on magnetic resonance contrast agents
* Patients with a Decreased renal function(Glomerular filtration rate <30 mL / min)
* Other, maternity, patients with a pacemaker or a cochlear

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
pattern of lymph drainage (Scale of 0 to 5) | After magnetic resonance lymphangiography scans in up to 2years
  0(abnormal)-10(normal)
delay of lymph drainage (Scale of 0 to 10) | After magnetic resonance lymphangiography scans in up to 2years
  0(delay)-10(normal)
depiction of lymph vessels (Scale of 0 to 10) | After magnetic resonance lymphangiography scans in up to 2years
  0(Not clarity)-10(Clarity)
enhancement of inguinal lymph nodes (Scale of 0 to 10) | After magnetic resonance lymphangiography scans in up to 2years
  0(Not clarity)-10(Clarity)
Visibility of Lymphatic Duct (Scale of 0 to 10) | After magnetic resonance lymphangiography scans in up to 2years
  0(Invisible)-10(Clearly visible)

CONTACTS AND LOCATIONS:
Overall Officials: SeungHong Choi, MD,PhD, Principal Investigator — Seoul National University Hospital(Radiology)
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea